CLINICAL TRIAL: NCT02335398
Title: Development and Evaluation of a Methadone Protocol for Severe Chronic Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 289/2554(EC4)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Pain, Chronic
Keywords: methadone; chronic pain; noncancer pain; cancer pain; QTc prolongation
MeSH Terms: conditions — Chronic Pain; Cancer Pain | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- methadone (Experimental): single group
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — The starting methadone dose for naïve-opioid patients was 2.5-5 mg every 8-12 hours. In patients who required opioid rotation, the conversion ratios, morphine:methadone, were 4:1, 8:1, and 12:1 for patients receiving less than 90 mg of morphine, receiving 90-300 mg of morphine, and receiving more than 300 mg of morphine , respectively. A fixed dose ratio of 1:20 was applied for changing from transdermal fentanyl to oral methadone. Then, the daily calculated methadone dose was divided into 8-12 hourly dosing. Calculated rescue dose was estimated to be 10-15% of total daily dose of methadone which there was switched to be morphine syrup in the ratio of 1:4.
  Other Names: Methadone GPO

SUMMARY:
Methadone is a synthetic mu opioid agonist that has been proved as clinically effective in pain management. However, methadone usage for pain control in Thailand has been limited because physicians are not familiar with its dosing and concern about the risk of drug accumulation and cardiac arrhythmia. Therefore, this prospective study was conducted to evaluate the efficacy and safety of a methadone protocol in Thai patients with severe chronic noncancer and cancer pain.

DETAILED DESCRIPTION:
Chronic pain is defined as pain that persists beyond normal tissue healing time, which is assumed for 3 months by the IASP. The symptoms include either continuous or intermittent pain, that could be caused by tumor or other multiple etiologies. The consequence of uncontrolled chronic pain presents not only physiologic symptoms but also psychiatric disorders leading to severely impact daily living.

In Thailand, the use of methadone for pain management has been limited because physicians are not familiar with its dosing and concern about the risk of drug accumulation and cardiac arrhythmia. Therefore, the aim of this study is to evaluate the efficacy and safety of a protocol of methadone dosing in outpatients with severe chronic pain.

Thirty four chronic pain patients will be included to initiate methadone use following the protocol. Pain scores, pain interferences scores, neuropathic pain score, severity of adverse effects, and QTc intervals will be assessed at baseline, and two, four, eight, and twelve weeks after starting methadone.

The approved protocol of methadone therapy obtained from this study could be clinically utilized by physicians for severe chronic pain management.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 or over who suffered from severe chronic cancer or noncancer pain to be firstly treated with methadone as analgesics

Exclusion Criteria:

* QTc interval that was more than 500 msec
* History of opioid addiction
* Having structural heart diseases
* During pregnancy or lactation period
* Patients who have hypersensitivity to methadone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain score | 3 months
  pain scores are assessed at baseline, and two, four, eight, and twelve weeks after starting methadone.

SECONDARY OUTCOMES:
pain interferences scores | 3 months
  pain interferences scores are assessed at baseline, and two, four, eight, and twelve weeks after starting methadone.
severity of adverse effects | 3 months
  severity of adverse effects are assessed at baseline, and two, four, eight, and twelve weeks after starting methadone
QTc intervals | 3 months
  QTc intervals are assessed at baseline, and two, four, eight, and twelve weeks after starting methadone
Neuropathic pain score | 3 months
  Neuropathic pain score are assessed at baseline, and two, four, eight, and twelve weeks after starting methadone

CONTACTS AND LOCATIONS:
Overall Officials: Chuthamanee Suthisisang, Ph.D., Study Chair — Thailand: Faculty of Pharmacy, Mahidol University; Phutsadee Pudchakan, Bsc.Pharm, Principal Investigator — Thailand: Faculty of Pharmacy, Mahidol University; Krittika Tanyasaensook, Ph.D., Study Director — Thailand: Faculty of Pharmacy, Mahidol University; Pongparadee Chaudakshetrin, M.D., Study Director — Thailand: Faculty of Medicine Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Mercadante S, Casuccio A, Calderone L. Rapid switching from morphine to methadone in cancer patients with poor response to morphine. J Clin Oncol. 1999 Oct;17(10):3307-12. doi: 10.1200/JCO.1999.17.10.3307. PMID 10506634
- [Background] Mercadante S, Casuccio A, Fulfaro F, Groff L, Boffi R, Villari P, Gebbia V, Ripamonti C. Switching from morphine to methadone to improve analgesia and tolerability in cancer patients: a prospective study. J Clin Oncol. 2001 Jun 1;19(11):2898-904. doi: 10.1200/JCO.2001.19.11.2898. PMID 11387363
- [Background] Ripamonti C, Groff L, Brunelli C, Polastri D, Stavrakis A, De Conno F. Switching from morphine to oral methadone in treating cancer pain: what is the equianalgesic dose ratio? J Clin Oncol. 1998 Oct;16(10):3216-21. doi: 10.1200/JCO.1998.16.10.3216. PMID 9779694
- [Background] Bruera E, Sweeney C. Methadone use in cancer patients with pain: a review. J Palliat Med. 2002 Feb;5(1):127-38. doi: 10.1089/10966210252785097. PMID 11839235
- [Background] Pearson EC, Woosley RL. QT prolongation and torsades de pointes among methadone users: reports to the FDA spontaneous reporting system. Pharmacoepidemiol Drug Saf. 2005 Nov;14(11):747-53. doi: 10.1002/pds.1112. PMID 15918160